CLINICAL TRIAL: NCT01840124
Title: Uterine Leiomyoma Treatment With Radiofrequency Ablation
Acronym: ULTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Davis (Other); University of California, Irvine (Other); University of California, Los Angeles (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-11026
Record Dates: First submitted 2013-04-17; First posted 2013-04-25 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Uterine Fibroids
Keywords: Fibroids; Radiofrequency ablation
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acessa (Experimental): All women in the trial will be in this group who receive treatment using the Acessa device.
  Interventions: Procedure: Radiofrequency ablation of fibroids

INTERVENTIONS:
Procedure: Radiofrequency ablation of fibroids — The Acessa device delivers radiofrequency energy to uterine fibroids to destroy fibroid tissue. The patient undergoes a standard laparoscopy of the pelvis. A laparoscopic ultrasound is performed to identify the precise size and location of the fibroids. The Acessa radiofrequency probe is then placed into the fibroid and the radiofrequency energy is delivered. The fibroid tissue is destroyed and the fibroid shrinks down in size to decrease fibroid-related symptoms.
  Other Names: Acessa

SUMMARY:
The ULTRA study is a single-arm trial of 100 premenopausal women with symptomatic uterine fibroids who undergo treatment with the Acessa device. The Acessa device is a new FDA approved minimally invasive treatment for uterine fibroids that uses radiofrequency energy to destroy fibroid tissue. The fibroids then shrink and symptoms are significantly improved. The radiofrequency energy is delivered to the fibroids during an outpatient surgical procedure. There is minimal blood loss and pain and women return to the usual activities 5-9 days after the Acessa procedure.

The investigators will evaluate changes in fibroid-related symptoms from before the Acessa treatment to 3, 6, 12, 18, 24, 30, and 36 months after Acessa treatment. The investigators will also assess operative outcomes including procedure duration, complications, blood loss, post-operative pain, and the time to return to usual activities. The investigators will determine long-term efficacy of Acessa by evaluating the rate of re-treatment for symptomatic fibroids after the Acessa procedure.

Study participants will be recruited at 5 sites within the UC Fibroid Network: UC Davis, UC Irvine, UC Los Angeles, UC San Diego, and UC San Francisco. UC San Francisco will serve as the Coordinating Center for the trial with oversight of all scientific and administrative aspects of the study. All study data will be stored securely in a HIPAA compliant, secure database monitored by the UC San Francisco Coordinating Center. A data safety and monitoring board will oversee participant safety and protection.

ELIGIBILITY:
INCLUSION CRITERIA

1. Premenopausal (at least 1 menstrual period in last 3 months)
2. Age >21years
3. Fibroids are associated with heavy bleeding, pelvic pressure or discomfort, urinary or bowel symptoms, or dyspareunia
4. Desires surgical management of fibroids
5. Uterus ≤16 weeks in size
6. All fibroids ≤ 10cm in maximum diameter by ultrasound or MRI assessment within the last year.
7. Total number of fibroids ≤6 by ultrasound or MRI assessment within the last year. (For this study "Fibroids" will be leiomyomas > 2cm)
8. Had a Pap smear within the last 3 years with appropriate follow-up and treatment for cellular abnormalities
9. Endometrial biopsy indicates no hyperplasia or cancer (biopsy only required if age >45 years and has anovulatory heavy bleeding)
10. Able to tolerate laparoscopic surgery
11. Able to give informed consent

EXCLUSION CRITERIA

1. Planned treatment for infertility
2. Pedunculated fibroid with thin stalk (total stalk length is <25% maximum diameter of fibroid)
3. Intracavitary (FIGO Type 0) fibroid
4. Symptomatic fibroids are only FIGO Type 1 (submucosal with ≥ 50% intracavitary)
5. Planned concomitant surgical procedure in addition to treatment of uterine fibroids
6. Use of Essure or any other metallic, implantable device within pelvis
7. Pregnancy
8. Pelvic infection with the last 3 months
9. History of pelvic malignancy and/or pelvic radiation
10. Known or high suspicion for dense pelvic adhesions
11. Fibroids treated by myomectomy, uterine artery embolism, radio-frequency ablation, MRI Guided focused ultrasound, or cryomyolysis within the last 3 months

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Changes in fibroid-related symptoms after the Acessa procedure. | Baseline to 3 years.
  Changes as assessed by standard questionnaires for fibroid symptoms including menstrual pattern and flow and overall quality of life.

SECONDARY OUTCOMES:
Re-intervention for recurrent fibroid symptoms following the Acessa procedure. | Baseline to 3 years
Operative complications | Baseline to 6 weeks
  Operative complications are rare but may include excessive blood loss, uterine or pelvic infection, injury to organs adjacent to uterus such as bowel or bladder.
Pregnancy after the Acessa procedure | Baseline to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Jacoby, MD, Principal Investigator — University of California, San Francisco
Locations (5):
- United States (5):
  - University of California, Davis, Davis, California
  - University of California, Irivine, Irvine, California
  - University of California, San Diego, La Jolla, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California

REFERENCES:
- See also: Fibroid Trials at UCSF — https://clinicaltrials.ucsf.edu/fibroids

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT01840124/Prot_SAP_000.pdf